CLINICAL TRIAL: NCT02473562
Title: Varenicline, a Partial Nicotinic Receptor Agonist for the Treatment of Excessive Daytime Sleepiness in Parkinson's Disease: a Placebo-controlled Cross-over Pilot Study
Brief Title: Varenicline Treatment for Excessive Daytime Sleepiness in Parkinson's Disease
Acronym: VESPA
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: insufficient patient enrollment, insufficient funds for completion
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Centre for Human Drug Research, Netherlands (Other)
Responsible Party: Principal Investigator, Tom van Mierlo, MD, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NL40128.029.12
Record Dates: First submitted 2015-06-12; First posted 2015-06-16 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Varenicline; Excessive daytime sleepiness
MeSH Terms: conditions — Parkinson Disease; Disorders of Excessive Somnolence | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Varenicline (Experimental): Varenicline capsule 1 mg BID
  Interventions: Drug: Varenicline
- Placebo (Placebo Comparator): Placebo capsule
  Interventions: Drug: Placebo (for varenicline)

INTERVENTIONS:
Drug: Varenicline — Tablet 1 mg BID
  Other Names: Champix
  Arms: Varenicline
Drug: Placebo (for varenicline) — Tablet 1 mg BID
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The effect of varenicline, an alpha4beta2 nicotinic receptor partial agonist on excessive daytime sleepiness in Parkinson's disease will be studied in a randomized, double blind, placebo-controlled clinical trial with a within-subject crossover design.

DETAILED DESCRIPTION:
Sleep disturbances are common in Parkinson's disease and include excessive daytime sleepiness that has been reported in up to 50% of patients. Relatively little therapeutic research has addressed the problem of excessive daytime sleepiness and current treatment is largely aimed at reducing the dose of dopaminergic medication while trying to maintain sufficient motor control which unfortunately often fails. Apart from degeneration of dopaminergic neurons, a decrease in cholinergic projections to the brain arousal areas may be at least partly responsible for the occurrence of excessive daytime sleepiness in Parkinson's disease. Smoking in narcoleptic patients diminishes sleep attacks and excessive daytime sleepiness , thus one may hypothesize that nicotinergic stimulation of the brain arousal areas may improve excessive daytime sleepiness in Parkinson's disease. Therefore the effect of varenicline, an alpha4beta2 nicotinic receptor partial agonist, on excessive daytime sleepiness in Parkinson's disease will be studied in a placebo-controlled cross-over study.

ELIGIBILITY:
Inclusion Criteria:

* idiopathic Parkinson's Disease according to clinical diagnostic criteria United Kingdom Parkinson's Disease Society Brain Bank
* receiving stable Parkinson's medications for at least four weeks before and throughout study
* suffering Excessive Daytime Sleepiness, defined by a score of >10 on the Epworth Sleeping Scale
* written informed consent

Exclusion Criteria:

* Parkinson's Disease patients receiving medications with known central depressant effects (benzodiazepines, neuroleptics, anticholinergics)
* dementia defined by a Mini Mental State Examination <24
* depression defined by a Beck Depression Inventory >16
* a known diagnosis of sleep apnea or narcolepsy
* current smoking or smoking cessation in past 6 months
* presence of contra-indications for treatment with varenicline, including:

  * known psychiatric diseases such as panic disorder, psychosis, bipolar disorder, eating disorder and alcohol or drug abuse
  * unstable angina, a history of cardiac disease or stroke in previous 6 months
  * severe renal failure (glomerular filtration rate ≤ 30 ml/min)
  * insulin-dependent diabetes

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Daytime sleepiness | 4 weeks
  Epworth Sleepiness Scale

SECONDARY OUTCOMES:
Sleep quality | 4 weeks
  Pittsburgh Sleep Quality Index
Fatigue | 4 weeks
  Fatigue Severity Scale
Involuntary movements | 4 weeks
  Abnormal Involuntary Movements Scale
Quality of life | 4 weeks
  Medical Outcomes Study 36-Item Short-Form Health Survey
Sleep latency | 4 weeks
  Maintenance of Wakefulness Test
Pharmacodynamics assessed by computerized test battery | 4 weeks
Error score | 4 weeks
  Sustained Attention to Response Test

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Foncke, PhD, MD, Study Chair — VU University Medical Center, depart. of neurology; Bernard Uitdehaag, Phd, MD, Principal Investigator — VU University Medical Center, depart. of neurology; Tom van Mierlo, MD, Study Director — VU University Medical Center, depart. of neurology
Locations (2):
- Netherlands (2):
  - Academic Medical Center, Amsterdam
  - VU university medical center, Amsterdam